CLINICAL TRIAL: NCT03744130
Title: Contrast-enhanced Bowel Ultrasound in Making a Diagnosis and Follow-up of Patients With Inflammatory Bowel Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: State Scientific Centre of Coloproctology, Russian Federation (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 34A
Record Dates: First submitted 2018-11-14; First posted 2018-11-16 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Inflammatory Bowel Disease
Keywords: Contrast-enhanced Ultrasound; Inflammatory Bowel Disease; CD; UC; SonoVue; Endoscopic activity
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- patients with UC (Experimental): Patients with endoscopically proven UC with various extents of disease activity.
  Diagnostic Test: Contrast-enhanced Ultrasound
  Interventions: Diagnostic Test: Contrast-enhanced Ultrasound
- patients with CD (Experimental): Patients with proven CD with various extents of disease activity Diagnostic Test: Contrast-enhanced Ultrasound
  Interventions: Diagnostic Test: Contrast-enhanced Ultrasound

INTERVENTIONS:
Diagnostic Test: Contrast-enhanced Ultrasound — 1. administration of drotaverine hydrochloride (No-Spa ®) to reduse excessive peristaltic movement
  2. visualization of the previously chosen affected bowel segment with the use of DCE-US (Dynamic Contrast-Enhanced Ultrasound) technology
  3. administration of 2.4 ml SonoVue® intravenously with a bolus injection through a peripheric venous line (left antecubital vein), followed by a 10ml 0.9% Natrium Chloride bolus
  4. the video-loop is acquired during contrast agent administration and wash-out (preferable loop duration - 3 min)
  5. the original DICOM loop is sent to a work station

SUMMARY:
The purpose of this study is to determine the efficacy of SonoVue® in participants with Crohn's disease and ulcerative colitis to various aspects including type of Inflammatory Bowel Disease, disease activity, the need for surgical treatment.

DETAILED DESCRIPTION:
Each patient is subjected to clinical, laboratory and endoscopic evaluation, each eligible patient is assigned to one of the arms:

Arm 1: patients with ulcerative colitis (50 patients) Arm 2: patients with Crohn's disease (50 patients) In each arm, patients are classified according to clinical an endoscopic activity of the disease.

Each patient is subjected to ultrasound examination of the bowel using a Philips iU 22 machine according to a standardized protocol:

* 12h fasting period
* exploratory scanning with the use of convex C5-1 probe
* detailed scanning with the use of linear L 12-5 probe with Power Doppler
* choosing a bowel segment with the most prominent changes
* Contrast-enhanced Ultrasound (CEUS)

CEUS is performed according to the following protocol:

* administration of drotaverine hydrochloride (No-Spa ®) to reduse excessive peristaltic movement
* visualization of the previously chosen affected bowel segment with the use of DCE-US (Dynamic Contrast-Enhanced Ultrasound) technology
* administration of 2.4 ml SonoVue® intravenously with a bolus injection through a peripheric venous line (left antecubital vein), followed by a 10ml 0.9% Natrium Chloride bolus
* the video-loop is acquired during contrast agent administration and wash-out (preferable loop duration - 3 min)
* the original DICOM loop is sent to a work station Philips QLab platform is used to acquire a fitted Local Density Random Walk Wash-in Wash-out algorithm (LDRWIWO algorhithm) time-intensity curve of contrast agent wash-in and wash-out. Qualitative and quantitative (Time to peak, Rise time, Mean transit time, Wash-in Slope, Peak intensity, Area under curve, Time from peak to one half) parameters are calculated for each region of interest (ROI).

ELIGIBILITY:
Inclusion Criteria:

* patient with verified UC/CD aged from 18 to 60y
* signed informed consent form for the study

Exclusion Criteria:

* pregnancy
* known allergy or history of adverse reaction to sulfur hexafluoride preparations
* marked pulmonary hypertension
* uncontrolled hypertension

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-01-10 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Correlation between contrast-enhanced ultrasound time-intensity curves and endoscopic disease activity | [7 days]
  Particular time-intensity curve characteristics (AUC, Peak intensity etc.) could correlate with endoscopic activity of ulcerative colitis

SECONDARY OUTCOMES:
Correlation between contrast-enhanced ultrasound time-intensity curves in patients with Crohn disease and fibrosis grade according to morphologic analysis of the resected bowel segment | [14 days]
  Particular time-intensity curve characteristics could correlate with grade of fibrosis in the resected bowel segment

CONTACTS AND LOCATIONS:
Overall Officials: Larisa P Orlova, M.D., Principal Investigator — State Scientific Centre of Coloproctology, Russian Federation
Locations (1):
- State Scientific Centre of Coloproctology, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No